CLINICAL TRIAL: NCT04978909
Title: The Effectiveness of Tidal Volume Challenge Incorporating Plethysmographic Variability Index in Predicting Fluid Responsiveness
Brief Title: PVI for TVC Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202104002RINC
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Validation of PVI in Tidal Volume Challenge Test
Keywords: tidal volume challenge,Plethysmography variability index,Fluid responsiveness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine the ability of changes in Plethysmographic Variability Index during tidal volume challenge to predict fluid responsiveness

DETAILED DESCRIPTION:
The change of Plethysmographic Variability Index after tidal volume challenge as a predictor of fluid responsiveness, confirmed with the change of SVV using Flotrac advance cardiac output monitor.

To determine whether the patient is fluid responder, Fluid challenge will be performed afterwards to confirm the patient's fluid responsiveness.

We also aim to calculate the least significant change for Plethysmographic Variability Index and Philips PPV system.

ELIGIBILITY:
Inclusion:

Patients undergoing elective major surgery (estimated > 2-hr) with general anesthesia and mechanical ventilation in supine position

Exclusion:

1. BMI < 18.5 or >30 kg/m2
2. Pregnant patient
3. Allergy to starch solution
4. estimated glomerular filtration rate< 60

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major surgery (estimated > 2-hr) with general anesthesia and mechanical ventilation in supine position
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The predictive ability of change in Plethysmographic Variability Index after Tidal volume challenge to predict fluid responsiveness | 20 minutes
  The change in value of Plethysmographic Variability Index after increasing VTE from 6 ml/kg to 8 ml/kg.

SECONDARY OUTCOMES:
Least significant change for Massimo PVI and Philips PPV | 20 minutes
  Calculate the least significant change for Massimo PVI and Philips PPV using data acquired from our electronic system

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan